CLINICAL TRIAL: NCT02175472
Title: Sixty Minute Exposure of Specific Bandwidth Light for the Treatment of Idiopathic Parkinson's Disease
Brief Title: Efficacy Study of Light Therapy as an Adjunctive Treatment for Parkinson's Disease
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: PhotoPharmics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CT1301
Record Dates: First submitted 2014-06-24; First posted 2014-06-26 (Estimated); Results first posted 2018-10-23 (Actual); Last update posted 2018-10-23 (Actual); Status verified 2018-10

CONDITIONS: Parkinson Disease
Keywords: Parkinson's disease; Light therapy; Circadian rhythm
MeSH Terms: conditions — Parkinson Disease

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Spectramax light therapy device (Active Comparator): Light therapy device which emits a specific bandwidth combination and intensity of light.
  Interventions: Device: Spectramax light therapy device
- Control light device (Sham Comparator): Light therapy device, identical in appearance and operation to the Spectramax device, except that it produces a different bandwidth and intensity, which is not believed to produce a therapeutic response.
  Interventions: Device: Control light device

INTERVENTIONS:
Device: Spectramax light therapy device — Spectramax light therapy device emits a specific combination of bandwidths and intensities of light.
  Arms: Spectramax light therapy device
Device: Control light device — The control light device is identical in appearance to the Spectramax light therapy device, except that when turned on, emits a different combination of bandwidths and intensity, not believed to produce a therapeutic response.
  Arms: Control light device

SUMMARY:
Light treatment was originally employed in Parkinson's disease (PD) to determine if it might be effective in treating co-existing symptoms of depression and insomnia. However, a preliminary double-blind study as well as other studies reported significant improvement in both motor and co-existing Parkinsonian symptoms. As of yet, no long term double blind study has validated these findings. This study will use a double-blind design to evaluate the safety and efficacy of a non-invasive light therapy device to be used with ongoing pharmacotherapy for PD, over a six month treatment period.

DETAILED DESCRIPTION:
Parkinson's disease (PD) is traditionally described as a disorder of compromised dopamine (DA) function in the nigro-striatal dopamine (NSD) system. This system extends from the midbrain, through the hypothalamus and into the forebrain to critical areas involved in the control of motor performance. Restoration of DA content in this system by administering the DA precursor L-dopa or DA agonists reinstates motor control, but provides only symptomatic relief with waning efficacy as the disease advances. Symptoms of depression and sleep disturbances are also commonly seen in PD patients, and the manifestation of these symptoms suggests impaired circadian function.

Although the involvement of the circadian system in PD was intimated in the first formal account of the disorder provided by James Parkinson, it was not until recently that circadian malfunction has been specifically cited as playing a major role in the development and progression of the disease. In addition to scattered reports depicting circadian-like features of PD and related syndromes, a large body of evidence describes the benefits of light therapy in PD from both the preclinical and clinical perspectives.

While the development of a formal understanding has been largely omitted as to the basis for any therapeutic effect exerted by light, recent studies have shown that the nigro-striatal dopamine system is comprised of the same cell type as cells in the retina and the pineal. Such cells are driven by visual input whereby dopamine and melatonin sit in functional opposition to regulate day night activities including sleep, mood, reproduction, anti-oxidation and movement. Hence one may conclude that the circadian system plays a major role in many aspects of PD.

Recent work in PD has also suggested that the efficacy of light therapy is mediated by melatonin and dopamine function in the retina. On this basis it would be reasonable to assume that intervention into the function of the circadian system with light therapy in PD patients might well serve to modify the course and consequences of the disease. The present study serves to extend this finding to the point of providing a practical, non-invasive method for helping patients.

ELIGIBILITY:
Inclusion Criteria:

* 1.Males and females, with Stage II - III, idiopathic Parkinson's disease, as assessed by Hoehn-Yahr Scale
* 2. On an optimized, stable dopamine replacement therapy for at least 1 month

Exclusion Criteria:

* 1. Participants younger than 45 years old
* 2. Participation in a study of investigational or marketed drugs or devices during the 30-day period prior to the prospective subject's Baseline Evaluation or during their involvement in this investigation
* 3. Subjects who are medically complicated, medically unstable and/or have other severe co-morbid disease states, as determined by the Investigator.
* 4. History of psychiatric illness that would preclude compliance with the protocol and/or ability to complete the study safely
* 5. History or current diagnosis of major psychiatric disorder including Bipolar I Disorder that could interfere with accurate assessment and effective treatment
* 6. Have a Beck Depression Inventory-II (BDI-II) score of greater than or equal to 14
* 7. An anticipated need for a change in dopamine replacement therapy during the subject's involvement in the investigation
* 8. Patients on stable anti-depressant dose for less than 6 weeks
* 9. Less than one month since stopping an anti-depressant or psychoactive medication
* 10. History of current or recent (within previous 12 months) alcohol, narcotic or other drug abuse by the Diagnostic and Statistical Manual of Mental Disorders 5th Edition (DSM-5) criteria
* 11. Active suicidal or homicidal ideation or plan as determined by the Investigator or have a score of greater than or equal to 2 on the DBDI-II.
* 12. Previous use of light therapy treatment
* 13. Females of childbearing potential, i.e. capable of becoming pregnant
* 14. Night shift work within the past 6 months or planned during the investigation
* 15. Have planned travel of more than two weeks outside of two time zones from home during involvement in the Investigation
* 16. Planned travel outside of two time zones from home during the last two months of the Subject's involvement in the Investigation
* 17. Current use or use within the previous 1 month of photosensitizing or other medications that in the opinion of the investigator would interfere with the safety of the Subject during the trial including

  * amiodarone
  * benoxaprofen
  * chlorpromazine
  * demeclocycline
  * fleroxacin
  * nalidixic acid
  * ofloxacin
  * piroxicam
  * porfimer
  * psoralens
  * quinidine
  * temoporfin tetracycline
  * oral isoretinoin (Accutane)
  * St. John's wort
  * melatonin
* 18. Have a history of significant eye trauma or disease, retinopathy, and/or cataract of a level that would significantly affect transmission or processing of light through either eye
* 19. Other neurological disorders that in the opinion of the Investigator would interfere with the conduct of the study
* 20. Pre-existing major joint problems that in the opinion of the Investigator would interfere with the conduct of the study
* 21. History of cerebral insult or central nervous system infection that in the opinion of the Investigator would preclude successful participation in Investigation related procedures
* 22. Cognitive impairment, e.g. as determined by the Montreal Cognitive Assessment, that in the opinion of the Investigator would interfere with the conduct of the Investigation
* 23. Focal neurological deficits that in the opinion of the Investigator would interfere with the conduct of the Investigation
* 24. High dopamine replacement therapy (DART) dosage levels or severe dyskinesia attributable to DART that would preclude successful participation in the Investigation related procedures or interventions in the opinion of the site Investigator

Min Age: 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 92 (Actual)
Dates: Start 2014-06; Primary Completion 2016-10 (Actual); Study Completion 2016-12-23 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Dan Adams, Study Director — PhotoPharmics, Inc.
Locations (3):
- United States (2):
  - Massachusetts General Hospital (MGH), Boston, Massachusetts
  - Aspen Clinical Research, Orem, Utah
- VU University Medical Center (VUmc), Amsterdam, MB, Netherlands

REFERENCES:
- [Derived] Wyman BT, Adams D, Hendrix S, Groves J, Croft W, Ellison N, Olanow CW, Kieburtz K. A double-blind, controlled trial of circadian effective light therapy in patients with Parkinson's disease. Neurotherapeutics. 2025 Oct;22(6):e00728. doi: 10.1016/j.neurot.2025.e00728. Epub 2025 Sep 2. PMID 40903343

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Spectramax Light Therapy Device | Control Light Device
Started | 45 | 47
Completed | 38 | 45
Not Completed | 7 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Spectramax Light Therapy Device | Control Light Device | Total
Number analyzed (Participants) | 45 | 47 | 92
Age, Continuous [Mean (Standard Deviation); unit: years] | 70.3 (7.94) | 65.9 (7.55) | 68.0 (8.01)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 12 | 17 | 29
  Male | 33 | 30 | 63
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 1 | 1
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 45 | 46 | 91
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  Netherlands | 15 | 15 | 30
  United States | 30 | 32 | 62

OUTCOME MEASURES:

1. Primary Outcome: Change in the Combined Scores (Sum) of Parts I, II, and III of the Movement Disorders Society-Unified Parkinson's Disease Rating Scale (M (MDS-UPDRS) From Baseline to Endpoint at 6 Months.
Description: Part I: Non-motor impact of experiences of daily living. Part I has 13 questions,the first 6 are assessed by the examiner, and the remaining 7 are usually self assessed, but may include the patient's caregiver. Each question = 0-4, range= 0 - 65.
  Part II: Motor Aspects of Experiences of Daily Living: This portion of the scale assesses the motor impact of PD on patients' experiences of daily living. There are 13 questions which are a component of the self-administered Patient Questionnaire.Each question = 0-4, range = 0-65.
  Part III: Motor Examination: This portion of the scale assesses the motor signs of PD and is administered by the evaluator. There are 18 questions, however several questions have multiple parts which are also scored. Each question 0-4, Total range=0-132. Higher score=more severe
Time Frame: Six Months
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Spectramax Light Therapy Device | Control Light Device
Number analyzed (Participants) | 44 | 47
units on a scale | -17.7 (2.8) | -9.7 (3.5)

2. Secondary Outcome: Change in the Clinical Global Impression- Improvement Scale (CGI-I) From Baseline to Endpoint at 6 Months.
Description: The Clinical Global Impression of Improvement is an assessment of the clinician's view of the patient's global functioning. Participants are ranked "O" at baseline. The CGI-I ranks 0 - 7, with "0" being much improved, "4" being neutral, and "7" being much worse.
Time Frame: Six months
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Spectramax Light Therapy Device | Control Light Device
Number analyzed (Participants) | 44 | 47
units on a scale | -0.6 (0.1) | -0.2 (0.1)

3. Secondary Outcome: Change in the Score of the Parkinson's Disease Questionnaire - 39 From Baseline to Endpoint at 6 Months
Description: The 39 question Parkinson's Disease Questionnaire (PDQ-39) is a widely used patient reported rating scale in Parkinson's disease. Respondents affirm if they have experienced problems due to their disease using a five point scale from never (0 points) to always (4 points, or worse) in doing common activities. The PDQ-39 is comprised of 8 domains: mobility, emotion, activities of daily living, cognition, stigma, social support, communication, bodily discomfort. Total possible range of scores = 0 - 156
  The questions are divided into eight measurement scales each comprising 3 to 10 questions. The scores for the questions in each scale are totaled and normalized to a scale of 0 - 100, that is equivalent to percent of maximum score. The scales are; Mobility (MOB): Q1-10; Activities of Daily Life (ADL): Q11-16; Emotional Well Being (EMO): Q17-22; Stigma (STI): Q23-26; Social Support (SOC): Q27-29; Cognitions (COG): Q30-33; Communication (COM) Q34-36; and Bodily Discomfort (BOD): Q37-39.
Time Frame: Six months
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Spectramax Light Therapy Device | Control Light Device
Number analyzed (Participants) | 44 | 47
units on a scale | -1.3 (2.1) | 4.3 (1.7)

4. Secondary Outcome: Change in the Score of the Parkinson's Disease Sleep Scale-Disturbed Sleep, From Baseline to Endpoint at 6 Months.
Description: The Parkinson's Disease Sleep Scale 2 (PDSS-2) is designed to assess nocturnal disability in Parkinson's disease. The PDSS-2 is a 15 question analog scale that ranks answers from 0 - 4, with 4 being worse. In addition to an overall assessment of sleep disability three aspects of sleep problems can be obtained; disturbed sleep (total of questions 1-3, 8 and 14), PD-specific nocturnal motor symptoms (total of questions 4-6, 12 and 13), and PD-specific nocturnal symptoms (Total of questions 7, 9-11 and 15). We selected the "Disturbed Sleep" subscale as a key secondary outcome measure. This subscale has a total range of 0 - 16, with 16 being more severe.
Time Frame: Six months
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Spectramax Light Therapy Device | Control Light Device
Number analyzed (Participants) | 44 | 47
units on a scale | -0.0 (0.6) | 0.7 (0.5)

5. Secondary Outcome: Change in the Score of the Epworth Sleepiness Scale From Baseline to Endpoint at 6 Months.
Description: The Epworth Sleepiness Scale (ESS) is a scale intended to measure daytime sleepiness to help in diagnosing sleep disorders. The ESS questionnaire asks the subject to rate his or her probability of falling asleep on a scale of increasing probability from 0 (none) to 3 (worse) for eight different everyday situations. The total range is 0 - 24, with higher scores representing worse severity.
Time Frame: Six months
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Spectramax Light Therapy Device | Control Light Device
Number analyzed (Participants) | 44 | 47
units on a scale | -1.4 (0.6) | 0.1 (0.5)

ADVERSE EVENTS:
Time Frame: Adverse events were collected from baseline through the endpoint at Month 6, as well as the follow-up Month 7. Because the baseine period also included a two week period, the total safety data collection period was 7.5 months.
Description: Adverse events were recorded in the following ways: During the bi-weekly phone calls made by the study coordinator to each patient, during patient evaluations, during post evaluation interviews, and if the patient called to report an adverse event. Participants were asked during the phone calls, evaluations and interviews to report any event.
Arm/Group | Spectramax Light Therapy Device | Control Light Device
Serious Adverse Events (participants affected / at risk) | 3/45 | 1/47
Other Adverse Events (participants affected / at risk) | 5/45 | 2/47
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Spectramax Light Therapy Device (N=45) | Control Light Device (N=47)
Transient Ischemic Attack (Cardiac disorders) | 1 (1) | 0 (0)
Hip deterioration (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) — Hip deterioration requiring surgery
Accident (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) — Subject hit by car while walking on sidewalk
Rib fracture (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) — Subject fell and broke 2 ribs
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Spectramax Light Therapy Device (N=45) | Control Light Device (N=47)
Eye disorders and other eye related problems (Eye disorders) | 5 (5) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other